CLINICAL TRIAL: NCT01040767
Title: Comparison of Web- Versus Classroom-based Basic Ultrasound and EFAST Training in Two European Hospitals
Brief Title: Comparison of Web- Versus Classroom-based Basic Ultrasound and Extended Focused Assessment With Sonography for Trauma (EFAST) Training in Two European Hospitals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Klinikum Nürnberg (Other); Institut fuer Notfallmedizin Kempten e.V., Germany (Unknown)
Responsible Party: Elke Platz, MD, RDMS, Department of Emergency Medicine, Brigham and Women's Hospital, Boston, USA
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2008-P-002019/1
Record Dates: First submitted 2009-12-24; First posted 2009-12-30 (Estimated); Last update posted 2009-12-30 (Estimated); Status verified 2009-12

CONDITIONS: Learning
Keywords: Ultrasound education; Blended learning; Distance education; Trauma ultrasound; FAST

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Class (Active Comparator)
  Interventions: Other: Didactic training in basic ultrasound and the EFAST
- Web (Active Comparator)
  Interventions: Other: Didactic training in basic ultrasound and the EFAST
- Control (No Intervention)

INTERVENTIONS:
Other: Didactic training in basic ultrasound and the EFAST — Physicians in the classroom group (class) listened to traditional lectures, while the web group (web) watched narrated lectures online. All participants completed a pre- and post-test, and a second post-test eight weeks later. Both groups underwent hands-on training after the first post-test.
  Arms: Class; Web

SUMMARY:
Study Objective: Training physicians in new skills via classroom-based teaching has inherent costs and time constraints. We sought to evaluate whether web-based didactics result in similar knowledge improvement and retention of basic ultrasound principles and the EFAST (Extended Focused Assessment with Sonography for Trauma) compared with the traditional method.

Methods: Physicians from two German emergency departments were randomized into a classroom group with traditional lectures and a web group that watched narrated lectures online. All participants completed a pre- and post-test, and a second post-test eight weeks later. Both groups underwent hands-on training after the first post-test. A control group completed the two initial tests without didactic intervention.

ELIGIBILITY:
Inclusion Criteria:

* Physicians currently practicing in a German emergency department
* Age ≥ 18 years

Exclusion Criteria:

* Inability to participate in all aspects of the study prior to study begin
* Control group: Subjects who did not complete the pre-test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Mean test scores by didactic group for three consecutive multiple choice tests | November 2008 - February 2009

SECONDARY OUTCOMES:
Participant satisfaction with training and reported comfort with ultrasound use after training | December 2008 - February 2009

CONTACTS AND LOCATIONS:
Overall Officials: Elke Platz, MD, RDMS, Principal Investigator — Brigham and Women's Hospital, Boston USA
Locations (2):
- Germany (2):
  - Institut fuer Notfallmedizin e.V., Kempten (Allgäu), Bavaria
  - Klinikum Nuernberg, Nuremberg, Bavaria